CLINICAL TRIAL: NCT02586948
Title: Physiological Study of Minimally Invasive Extracorporeal CO2 Removal in Exacerbations of COPD Requiring Invasive Mechanical Ventilation
Brief Title: Physiological Study of Minimally Invasive ECCO2R in Exacerbations of COPD Requiring Invasive Mechanical Ventilation
Acronym: EPHEBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Alung Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAO14044
Record Dates: First submitted 2015-08-31; First posted 2015-10-27 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: extracorporeal CO2 removal
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- extracorporeal CO2 removal (Experimental): extracorporeal CO2 removal initiated shortly after intubation, using the veno-venous Hemolung device
  Interventions: Device: extracorporeal CO2 removal (Hemolung device)

INTERVENTIONS:
Device: extracorporeal CO2 removal (Hemolung device) — ECCO2R in severe exacerbation of COPD patients, requiring invasive mechanical ventilation with persistent respiratory acidosis and dynamic hyperinflation
  Other Names: ECCO2R

SUMMARY:
Morbidity and mortality in COPD result largely of acute exacerbations.The optimization of the respiratory management represents a fundamental challenge for improving prognosis and reducing mortality. While the hospital mortality of patients treated with NIV has decreased over years, and is currently less than 10 %, mortality in patients treated with invasive ventilation remains higher than 25%. To improve the prognosis of patients with acute exacerbation of COPD requiring invasive mechanical ventilation is therefore a major challenge in terms of morbidity and mortality. Among the means available to achieve this goal, minimally invasive extracorporeal CO2 removal (ECCO2R) seems to be a very promising approach.

The investigators hypothesize that the addition of minimally invasive ECCO2R is likely to limit dynamic hyperinflation in COPD patients requiring invasive mechanical ventilation for an acute exacerbation, while improving gas exchange.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is currently the fourth leading cause of death in the U.S. and is expected to become the third leading cause of death in 2020. Morbidity and mortality in COPD result largely of acute exacerbations, which are responsible for 1.5 million ED visits and 750,000 hospitalizations per year in the U.S. The optimization of the respiratory management of acute exacerbations represents a fundamental challenge for improving prognosis and reducing mortality. The value of non-invasive ventilation (NIV) for severe acute exacerbations of COPD was formally demonstrated by randomized clinical trials. In the setting of severe COPD exacerbations, NIV is actually very largely employed, largely ahead from invasive mechanical ventilation. While the hospital mortality of patients treated with NIV has decreased over years, and is currently less than 10 %, mortality in patients treated with invasive ventilation remains as high than 25%. Mortality in patients treated with invasive ventilation after failure of NIV seems to be growing and is actually close to 30%. To improve the prognosis of patients with acute exacerbation of COPD requiring invasive mechanical ventilation is therefore a major challenge in terms of morbidity and mortality. Among the means available to achieve this goal, minimally invasive extracorporeal CO2 removal (ECCO2R) seems to be a very promising approach.

The investigators hypothesize that the addition of minimally invasive ECCO2R is likely to limit dynamic hyperinflation in COPD patients requiring invasive ventilation for an acute exacerbation, while improving gas exchange. If confirmed, it could imply a more rapid weaning from invasive ventilation in relation to:

* less hemodynamic consequences of positive pressure ventilation
* reduced risk of baro-volo trauma of the lung parenchyma
* reduction in the use of sedative drugs
* a chest configuration minimizing diaphragmatic flattening, therefore favoring the generation of higher trans-diaphragmatic pressures
* a decrease in the work of breathing (WOB), in connection with the previous point and with a decrease in alveolar ventilation required for pulmonary CO2 elimination during the ECCO2R treatment All of these elements are clinically relevant, as a reduction in the duration of invasive ventilation is associated in the literature with a decrease in the incidence of pneumonia associated with mechanical ventilation, as well as with a decrease in the duration of ICU-stay.

ELIGIBILITY:
Inclusion Criteria:

* clinical exacerbation of a known or suspected COPD
* intubation and invasive mechanical ventilation since less than 72 hrs.
* ACV or CV mode (VT 8 ml/kg, RR 12/min., PEEP : 0 cmH20)
* pH < 7.30 and PaCO2 > 55 mm Hg and PEEPi (end-expiratory occlusion) > 5 cmH20
* written inform consent (patient, patient's legal surrogate)
* affiliation to a social security regime

Exclusion Criteria:

* Body Mass Index (BMI) > 35 kg/m2
* PaO2/FiO2 < 200 mm Hg
* history of hemorrhagic stroke
* heparin-induced thrombocytopenia
* Severe thrombopenia type II history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07; Primary Completion 2018-01-14 (Actual); Study Completion 2018-02-12 (Actual)

PRIMARY OUTCOMES:
intrinsic PEEP (PEEPi) | 12 hours (between measurements at baseline and under ECCO2R)
  PEEPi at baseline and after ECCO2R by the Hemolung® device and adjustment of ventilator settings, expressed in cmH20

SECONDARY OUTCOMES:
Functional Residual capacity (FRC) | 12 hours (between measurements at baseline and under ECCO2R)
  FRC using the nitrogen washout method, expressed in mL
PaO2 | 12 hours (between measurements at baseline and under ECCO2R)
  PaO2 expressed in mmHg
PaCO2 | 12 hours (between measurements at baseline and under ECCO2R)
  PaCO2 expressed in mmHg
Arterial O2 saturation | 12 hours (between measurements at baseline and under ECCO2R)
  Arterial O2 saturation expressed in %
pH | 12 hours (between measurements at baseline and under ECCO2R)
  pH expressed in absolute value
amount of sedative drugs | Average time period of 6 days
  amount of sedative drugs (per day and cumulative)
length of intubation | Average time period of 7 days, up to 28 days
  length of intubation (days)
length of ICU-stay | Average time period of 8 days, up to 28 days
  length of ICU-stay (days)
length of hospital stay | Average time period of 9 days, up to 28 days
  length of hospital stay (days)
ICU mortality | Average time period of 9 days, up to 28 days
  Number of in ICU-deceased participants (expressed in absolute number and %)
catheter related complications | Average time period of 9 days
  catheter related complications (thrombosis, bleeding, pneumothorax, infection) expressed in total number of complications, in average number of complications per participant and in number of patients with complications
Hemolung related complications | Average time period of 9 days
  Hemolung related complications (thrombosis, bleeding) expressed in total number of complications, in average number of complications per participant and in number of patients with complications
non catheter-related bleedings | Average time period of 9 days
  non catheter-related bleedings expressed in total number of bleedings, in average number of bleedings per participant and in number of patients with bleedings
work of breathing per Liter | Average time period of 7 days
  work of breathing with and without ECCO2R, expressed in Joules per Liter of ventilation
work of breathing per minute | Average time period of 7 days
  work of breathing with and without ECCO2R, expressed in Joules per minute
work of breathing per breath | Average time period of 7 days
  work of breathing with and without ECCO2R, expressed in Joules per breath
Occlusion pressure in 100msec (P0.1) | Average time period of 7 days
  Occlusion pressure in 100msec in parallel to work breathing measurements with and without ECCO2, expressed in cmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Diehl, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - CHU d'Angers, Angers
  - Hopital de Bicetre, Hopitaux universitaires Paris Sud, Le Kremlin-Bicêtre
  - Hopital Europeen Georges Pompidou, Paris

REFERENCES:
- [Derived] Diehl JL, Piquilloud L, Vimpere D, Aissaoui N, Guerot E, Augy JL, Pierrot M, Hourton D, Arnoux A, Richard C, Mancebo J, Mercat A. Physiological effects of adding ECCO2R to invasive mechanical ventilation for COPD exacerbations. Ann Intensive Care. 2020 Sep 29;10(1):126. doi: 10.1186/s13613-020-00743-y. PMID 32990836